CLINICAL TRIAL: NCT03766607
Title: A Multi-center Phase II Study of Trastuzumab Biosimilar (SB3®) in Combination With Ramucirumab and Paclitaxel in HER2 Positive Metastatic Gastric Cancer Patients
Brief Title: Trastuzumab Beyond Progression in HER2 Positive Metastatic Gastric Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Competing other studies
Sponsor: Korean South West Oncology Group (Network)
Responsible Party: Principal Investigator, Hwan Jung Yun, Clinical Professor, Korean South West Oncology Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSWOG 1018
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab with Ramucirumab and Paclitaxel (Experimental): Single arm study of trastuzumab (8 mg/kg loading dose; 6 mg/kg maintenance) every 21 days + ramucirumab (8 mg/kg) on days 1 & 15 every 28 days + paclitaxel (80 mg/m2) on days 1, 8, and 15 every 28 days
  Interventions: Drug: Trastuzumab; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (8 mg/kg loading dose; 6 mg/kg maintenance) administered intravenously every 21 days
Drug: Ramucirumab — Ramucirumab 8 mg/kg administered intravenously on days 1 and 15 every 28 days
Drug: Paclitaxel — Paclitaxel 80 mg/m2 administered intravenously on days 1, 8, and 15 every 28 days

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of combination therapy with ramucirumab, paclitaxel, and trastuzumab biosimilar as second line treatment of HER2 positive metastatic gastric cancer after failure of first line chemotherapy including trastuzumab. This study is a phase II, single-arm, open label, multi-center study.

DETAILED DESCRIPTION:
Approximately 15% of patients with advanced gastric cancer have HER2 overexpression and the combined use of trastuzumab and other cytotoxic chemotherapeutic agents, such as 5-FU and cisplatin, in these patients is associated with a significantly improved survival rate compared with cytotoxic chemotherapy alone. So, the combination of trastuzumab and chemotherapy is currently being used as a standard treatment in HER2 positive advanced gastric or gastroesophageal adenocarcinoma. However, after failing first line treatment with such regimen, second line treatment is determined regardless of HER2 status, and the most preferred treatment is ramucirumab and paclitaxel combination chemotherapy.

Recently, the use of trastuzumab in combination with other cytotoxic chemotherapeutic agents has been reported to be superior to the use of cytotoxic chemotherapy alone in the treatment of patients with HER2 positive metastatic breast cancer. On the basis of several guidelines, it is recommended to extend the use of trastuzumab after disease progression. In addition, in some retrospective studies of metastatic gastric cancer, it has been reported that treatment with trastuzumab in combination with second line chemotherapy followed by first line chemotherapy including trastuzumab is beneficial and it is worthwhile to be tested in the prospective study. Furthermore, data on the safety and efficacy of cross-administration of trastuzumab biosimilar have not been available yet.

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Histologically confirmed HER2 overexpressing gastric cancer (HER2 overexpression is defined as IHC 3+ or FISH +)
3. Metastatic gastric cancer
4. Progressive disease has been confirmed after first line treatment including trastuzumab (If the recurrence occurred within 6 months after the completion of postoperative adjuvant therapy, it can be considered as first line treatment.)
5. At least one measurable or evaluable lesion according to RECIST ver 1.1
6. ECOG performance status 0 or 1
7. Appropriate major organ function as defined below, A. Absolute neutrophil count (ANC) ≥ 1,500/mm3 B. Platelet ≥ 100,000/mm3 C. Hemoglobin > 8.0 g/dL D. Total bilirubin ≤ 1.5 x ULN E. AST and ALT < 3 x ULN (if there is a live metastasis, AST and ALT ≤ 5 x ULN) F. Serum creatinine ≤ 1.5x ULN or CCr > 50 mL/min
8. Life expectancy is more than 12 weeks
9. Echocardiography at the time of enrollment showed an ejection fraction ≥ 50%
10. Previous adverse events of chemotherapy or radiotherapy has been resolved to less than grade 1 toxicity (exception: Alopecia, stable peripheral neuropathy, and manageable electrolyte imbalance by replacement therapy are acceptable if they are resolved to less than grade 2)
11. If the urine pregnancy test or serum beta-hCG result is negative in child bearing women
12. If the subject have signed the informed consent form approved by the IRB

Exclusion Criteria:

1. Symptomatic or unstable CNS metastasis (exception: appropriately treated brain metastasis without progression of more than 4 weeks after previous CT or MRI, and no steroid treatment for symptom relief is necessary)
2. Active virus, bacteria, or fungal infection (exception: HBV DNA titer is in the normal range for chronic hepatitis B carriers)
3. If previous chemotherapy or radiotherapy was applied within 3 weeks before the administration of study drug
4. If the subject has received major surgery within 4 weeks and the recovery is not complete before the administration of study drug
5. If there is a history of other malignancies within 3 years (exception: cervical intraepithelial cancer, well differentiated thyroid cancer, or skin cancer has been treated completely)
6. QTc interval > 480 msec, long or short QT syndrome, or Burgada syndrome. In addition, known prolongation of QTc interval or Torsade de Pointes
7. If there is a significant history of cardiovascular disease within 6 months, such as, myocardial infarction, unstable angina, significant cardiac arrhythmia, and uncontrolled hypertension (systolic BP > 180 mmHg, diastolic BP > 100 mmHg), congestive heart failure (NYHA class III-IV), pericardial effusion or pericardial tamponade, cardiomyopathy, cerebrovascular disease including transient ischemic stroke, and symptomatic pulmonary embolism.
8. History of symptomatic interstitial pneumonia
9. History of other psychiatric problems, abnormalities of laboratory test which have potential effects on administration of study drugs or participation on the study, or if the subject is inappropriate to be participated according to the investigator's decision (refusal to request and instruction, incooperative attitudes, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, PFS | up to 12 months
  as measured from the start of the treatment to the date of either documentation of disease progression or death

SECONDARY OUTCOMES:
Objective response rate, ORR | up to 6 months
  defined as the proportion of subjects who have a best overall response of complete response or partial response as assessed by RECIST 1.1
Overall survival, OS | up to 12 months
  defined as the time from the date of randomization until the date of death from any cause
Adverse event | up to 12 months
  as measured by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Kee Song, Principal Investigator — Korean Southwest Oncology Group
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No